CLINICAL TRIAL: NCT02084628
Title: Open-label, Multi-center Study to Evaluate the Safety, Efficacy, and Plasma Gadolinium Concentrations After an Intravenous Injection of 0.1 mL/kg Body Weight Eovist/Primovist for Enhanced Magnetic Resonance Imaging (MRI) of the Liver in Children 0 to 2 Months of Age
Brief Title: Magnetic Resonance Imaging of the Liver in Children 0-2 Months of Age With an Intravenous Injection of Eovist/Primovist Which is a Contrast Agent
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment discontinued due to rare medical condition in the age group 0 to 2 months
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16078; 2012-000952-32 (EudraCT Number)
Record Dates: First submitted 2014-02-06; First posted 2014-03-12 (Estimated); Results first posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-08

CONDITIONS: Magnetic Resonance Imaging
MeSH Terms: interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gadoxetate disodium (Eovist/Primovist, BAY86-4873) (Experimental): Participants to receive single dose of Eovist/Primovist as a manual injection at a dose of 0.1 milliliter per kilogram (mL/kg) body weight (BW) (0.025 millimole [mmol]/kg BW), followed by a flush of at least 5 mL saline (sodium chloride 0.9 percent [%] solution) manually.
  Interventions: Drug: Gadoxetate disodium (Eovist/Primovist, BAY86-4873)

INTERVENTIONS:
Drug: Gadoxetate disodium (Eovist/Primovist, BAY86-4873) — Participants to receive single dose of Eovist/Primovist as a manual injection at a dose of 0.1 milliliter per kilogram (mL/kg) body weight (BW) (0.025 millimole [mmol]/kg BW), followed by a flush of at least 5 mL saline (sodium chloride 0.9 percent [%] solution) manually.

SUMMARY:
This is an open-label, multi-center study involving babies 0-2 months of age who have liver problems (pathology) and need to have their liver and possibly, the bile ducts imaged using magnetic resonance imaging and injection of a contrast agent (dye). This agent is called Eovist. It has been marketed since 2004 and used in many countries all over the world.

The baby will have blood tests before and after the imaging is done to make sure that there are no unexpected findings before and after the imaging. Also 3 blood samples up to 8 hours after the injection will be obtained in order to measure how much of the dye is in the blood. The baby will have an intravenous line which can be used for the blood samples and will not need to be stick for the blood samples. Several radiologists will evaluate the images. The family doctor will be contacted to find out what was the diagnosis and treatment after the results of the MRI were known. Six months after the study, the parent(s)/legal guardian(s) will be contacted to make sure the that baby did not have any problems, especially with the skin, joints and eyes.

DETAILED DESCRIPTION:
In order to minimize bias in assessment of the images, blinded reading of the MR images will be performed by 2 blinded readers. The blinded readers will be independent board-certified pediatric radiologists who have no knowledge about the subjects and are not affiliated with any of the clinical sites.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-2 months (must be gestational age 37 to 41 weeks)
* Scheduled to undergo routine contrast-enhanced liver MRI
* Able to comly with the study procedures

Exclusion Criteria:

* Scheduled for any intervention (except lumbar puncture and bone marrow aspiration) during the study period
* If receiving chemotherapy, may have a change in treatment during the study period
* Contraindication for MRI
* Renal insufficiency (estimated glomerular filtration rate < 80% of age-adjusted normal mean value using the Schwartz formula)
* Acute renal failure
* Clinically relevant abnormal laboratory parameter, ie, greater than 3 times the upper limit of the normal range, in particular, liver enzymes and renal function. (Note: if elevations in liver enzyme levels are consistent with the underlying hepatobiliary disease, then the subject may be enrolled.)

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- United States (9):
  - Los Angeles, California
  - Palo Alto, California
  - Washington D.C., District of Columbia
  - Brooklyn, New York
  - New York, New York
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Seattle, Washington
  - Madison, Wisconsin

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — https://www.clinicaltrialsregister.eu/ctr-search/search

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 9 centres in United States of America (USA) and only one participant was recruited in one centre, between 13 February 2015 (first subject first visit) and 11 August 2015 (Last subject last visit).
Pre-assignment Details: One participant was enrolled in the study.
Groups:
- Gadoxetate Disodium (Eovist/Primovist, BAY86-4873): Participant to receive single dose of Eovist/Primovist as a manual injection at a dose of 0.1 milliliter per kilogram (mL/kg) body weight (BW) (0.025 millimole [mmol]/kg BW), followed by a flush of at least 5 mL saline (sodium chloride 0.9 percent [%] solution) manually.
Period: Overall Study
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Additional Diagnostic Information From Combined (Pre-contrast And Post-contrast) Images Compared With Pre-contrast Images
Description: Additional diagnostic information such as better delineation of the border of the lesion, better definition of the internal morphology of the lesion, better characterization of the lesion, better definition of the location of the lesion, better assessment of the communication of the lesion with respect to the biliary system obtained from the combined magnetic resonance (MR) images compared with pre-contrast MR images. Number of subjects with additional diagnostic information were recorded and analyzed.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Measure: Number; unit: participants
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Number analyzed (Participants) | 1
participants | 0

2. Primary Outcome: Number of Subjects With Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence that is, any unfavorable and unintended sign (including abnormal laboratory findings), symptom or disease in a subject or clinical investigation subject after providing written informed consent for participation in the study.
Time Frame: From the signing of the informed consent form until the 6 month post MRI follow-up
Measure: Number; unit: participants
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Number analyzed (Participants) | 1
participants | 0

3. Primary Outcome: Number of Subjects With Serious Adverse Events
Description: An serious adverse events (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From the signing of the informed consent form until the 6 month post MRI follow-up
Measure: Number; unit: participants
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Number analyzed (Participants) | 1
participants | 0

4. Secondary Outcome: Number of Lesions Detected for the Pre-contrast Images
Time Frame: Images were taken pre-injection
Measure: Number; unit: number of lesions
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Number analyzed (Participants) | 1
number of lesions | 0

5. Secondary Outcome: Number of Lesions Detected for the Combined Images
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Measure: Number; unit: number of lesions
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Number analyzed (Participants) | 1
number of lesions | 0

6. Secondary Outcome: Contrast Enhancement of the Liver for the Combined Images Assessed by Yes or no Question
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Measure: Number; unit: number of responses
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Number analyzed (Participants) | 1
number of responses
  Yes | 1
  No | 0

7. Secondary Outcome: Contrast Enhancement of the Biliary System for the Combined Images Assessed by Yes or no Question
Description: Biliary system included
  1. Gall bladder
  2. Cystic duct
  3. Common bile duct
  4. Right main bile duct
  5. Left main bile duct
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Measure: Number; unit: number of responses
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Number analyzed (Participants) | 1
number of responses
  Yes | 1
  No | 0

8. Secondary Outcome: Visualization of the Biliary System for the Pre-contrast and Combined Images Assessed by Yes or no Question
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Measure: Number; unit: participants
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Number analyzed (Participants) | 1
participants
  Pre-contrast Images: Yes | 0
  Pre-contrast Images: No | 1
  Combined Images: Yes | 0
  Combined Images: No | 1

9. Secondary Outcome: Change in Diagnosis for the Combined Images Compared With Precontrast Images
Description: Diagnosis based on the pre-contrast images will be indicated. If there is a change in the diagnosis based on the combined images, then the combined images diagnosis will be recorded.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Measure: Number; unit: participants
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Number analyzed (Participants) | 1
participants | 0

10. Secondary Outcome: Diagnostic Confidence for the Pre-contrast and Combined Images Assessed by Yes or no Question
Description: Diagnostic confidence was classified as not confident (No), confident (Yes), very confident (Yes).
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Measure: Number; unit: number of responses
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Number analyzed (Participants) | 1
number of responses
  Pre-contrast Images: Very Confident-Yes | 0
  Pre-contrast Images: Confident-Yes | 0
  Pre-contrast Images: Not Confident-No | 1
  Combined Images: Very Confident-Yes | 1
  Combined Images: Confident-Yes | 0
  Combined Images: Not Confident-No | 0

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent form until the 6 month post MRI follow-up
Arm/Group | Gadoxetate Disodium (Eovist/Primovist, BAY86-4873)
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Primarily based on study 13729 along with supporting data the FDA revised Eovist labeling to remove any age restriction from indication and decided that there are no further pediatric data requested. Consequently, study was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No